CLINICAL TRIAL: NCT01216748
Title: Clinical Evidence of pH Dependent ß2 Adrenergic Transport Mechanisms in the Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Matthias Salathe, Professor of Medicine, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20070583; R01HL060644 (NIH)
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Results first posted 2014-12-17 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2014-11

CONDITIONS: Healthy Volunteers
Keywords: airway blood flow; albuterol; acidosis; alkalosis
MeSH Terms: conditions — Acidosis; Alkalosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- health life-time non smokers (Experimental): health lifetime non-smokers will be challenged with 4 respiratory maneuvers:quiet breathing, hypocapnic hyperventilation, hypercapnic hyperventilation, and eucapnic hyperventilation
  Interventions: Other: quiet breathing; Other: Hypocapnic Hyperventilation; Other: Hypercapnic Hyperventilation; Other: eucapnic hyperventilation

INTERVENTIONS:
Other: quiet breathing — Subjects were instructed to breath normally at room air.
Other: Hypocapnic Hyperventilation — hypocapnic hyperventilation, the subjects were instructed to breathe fast and deep until their end-tidal pCO2 fell to 30 mmHg, corresponding to a systemic pH increase of about 0.1 pH units.
Other: Hypercapnic Hyperventilation — For hypercapnic hyperventilation, a modification of a previously described procedure (15). While monitoring SaO2 using pulse oximetry and end-tidal CO2 by mass-spectrometry on a breath by breath basis, CO2 was bled into the inspired air to achieve an end-tidal pCO2 of at least 55 mmHg
Other: eucapnic hyperventilation — For eucapnic hyperventilation, the subjects were instructed to increase their ventilation to the highest level of ventilation recorded in the previous two hyperventilation maneuvers, while CO2 was bled into the inspired air to maintain end-tidal pCO2 at 40 mmHg.

SUMMARY:
The purpose of this study was to determine if airway pH has an effect on albuterol-induced vasodilation in the airway. Methods: Ten healthy volunteers performed the following respiratory maneuvers: quiet breathing, hypocapnic hyperventilation, hypercapnic hyperventilation, and eucapnic hyperventilation

DETAILED DESCRIPTION:
The lungs provide a unique absorptive surface for drug delivery. Many inhaled drugs are rapidly absorbed into the airway because of their lipophilic chemical characteristics. However, the majority of the currently used β2-adrenergic bronchodilators cannot freely diffuse across the epithelial cell membrane because of their transient or permanent positive charge at physiological pH. Inhaled albuterol, a β2-adrenergic agonist used widely for the treatment of obstructive airway disease, is charged positively in neutral or acidic conditions and thus requires active transport across the airway epithelium. Previous studies in the lab have shown that albuterol uptake into airway epithelia occurs via a pH sensitive cation transporter (OCTN2). The vasodilator response to an inhaled β2-adrenergic agonist could be an expression of epithelial cation transport. The investigators propose that the magnitude and duration of vasodilation in the airway caused by an inhaled hydrophilic β2-adrenergic agonist such as albuterol may be altered by changes in airway pH. The purpose of this protocol is to determine the effect of ASL pH on the response of Qaw to inhaled albuterol by manipulating airway pH through ventilatory maneuvers in health subjects: hyperventilation to raise pH and ventilation with CO2 bleed-in to lower pH.

ELIGIBILITY:
Inclusion Criteria:

* Lifetime non-smokers
* FEV1 > 80% predicted value and FEV1/FVC > 0.75

Exclusion Criteria:

* Cardiovascular disease or use of cardiovascular or vasoactive drugs;
* Lung disease or use of airway drugs (i.e. inhaled corticosteroids, β adrenergic agonists);
* Respiratory infection during the 4 weeks preceding the study
* Use of systemic glucocorticoids within 4 weeks of the study
* Pregnant or nursing females

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Salathe, Principal Investigator — University of Miami
Locations (1):
- Pulmonary Human Research Laboratory, University of Miami School of Medicine, Miami, Florida, United States

REFERENCES:
- [Background] Vaughan J, Ngamtrakulpanit L, Pajewski TN, Turner R, Nguyen TA, Smith A, Urban P, Hom S, Gaston B, Hunt J. Exhaled breath condensate pH is a robust and reproducible assay of airway acidity. Eur Respir J. 2003 Dec;22(6):889-94. doi: 10.1183/09031936.03.00038803. PMID 14680074
- [Background] Paget-Brown AO, Ngamtrakulpanit L, Smith A, Bunyan D, Hom S, Nguyen A, Hunt JF. Normative data for pH of exhaled breath condensate. Chest. 2006 Feb;129(2):426-430. doi: 10.1378/chest.129.2.426. PMID 16478862
- [Background] Horvath G, Schmid N, Fragoso MA, Schmid A, Conner GE, Salathe M, Wanner A. Epithelial organic cation transporters ensure pH-dependent drug absorption in the airway. Am J Respir Cell Mol Biol. 2007 Jan;36(1):53-60. doi: 10.1165/rcmb.2006-0230OC. Epub 2006 Aug 17. PMID 16917073
- [Derived] Cancado JE, Mendes ES, Arana J, Horvath G, Monzon ME, Salathe M, Wanner A. Effect of airway acidosis and alkalosis on airway vascular smooth muscle responsiveness to albuterol. BMC Pharmacol Toxicol. 2015 Apr 2;16:9. doi: 10.1186/s40360-015-0008-y. PMID 25889594

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: healthy lifetime non smokers were challenged with 4 respiratory manouvers: quiet breathing, hypocapnic hyperventilation, hypercapnic hyperventilation, and eucapnic hyperventilation in random order.
Period: Overall Study
Arm/Group | All Study Participants
Started | 10
Quiet Breathing | 10
Hypocapnic Hyperventilation | 10
Hypercapnic Hyperventilation | 10
Eucapnic Hyperventilation | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Controls: health-lifetime non-smokers were enrolled
Arm/Group | Controls
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 45 [23 to 54]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Changes in Airway Blood Flow After 180μg Albuterol by Inhalation (ΔQaw) vs Baseline
Description: Effect of airway pH on albuterol responsiveness as reflected by the change in airway blood flow after 180μg albuterol by inhalation (ΔQaw) vs baseline.
Time Frame: 15 minutes after albuterol inhalation
Measure: Mean (Standard Error); unit: changes from baseline in μl.min-1.ml-1
Groups:
- Health Controls: Health lifetime non smokers were recruited.
Arm/Group | Health Controls
Number analyzed (Participants) | 10
changes from baseline in μl.min-1.ml-1
  quiet breathing | 16.8 (1.9)
  eucapnic hyperventilation | 14.5 (2.4)
  hypocapnic hyperventilation | -0.2 (1.8)
  hypercapnic hyperventilation | 2.0 (1.5)

2. Secondary Outcome: Exhaled Breath Condensate (EBC) pH Variation
Description: EBC samples were collected at each respiratory maneuver by directing the subject's exhaled breath into a pre-cooled (-10C) tube for 10 min.
  pH was measured immediately after collection.
Time Frame: 10 minutes after each respiratory manouver.
Measure: Mean (Standard Error); unit: pH
Arm/Group | Health Controls
Number analyzed (Participants) | 10
pH
  quiet breathing | 6.39 (0.14)
  hypocapnic hyperventilation | 6.31 (0.08)
  hypercapnic hyperventilation | 6.59 (0.15)
  eucapnic hyperventilation | 5.88 (0.14)

ADVERSE EVENTS:
Arm/Group | Health Controls
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No